CLINICAL TRIAL: NCT00217386
Title: Therapy of Early Stage Myelodysplastic Syndrome (MDS) With ATG and Etanercept
Brief Title: Anti-Thymocyte Globulin and Etanercept in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Bart L. Scott, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Treatment
Other Study IDs: 1872.00; FHCRC-1872.00; CDR0000430702 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; atypical chronic myeloid leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Antilymphocyte Serum; Etanercept

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: etanercept

SUMMARY:
RATIONALE: Biological therapies, such as anti-thymocyte globulin and etanercept, may stimulate the immune system in different ways and stop cancer cells from growing. Giving anti-thymocyte globulin together with etanercept may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving anti-thymocyte globulin together with etanercept works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with low- or intermediate-1-risk myelodysplastic syndromes treated with anti-thymocyte globulin and etanercept.
* Correlate ex vivo and in vitro phenotypic, cytogenetic, and functional disease characteristics with in vivo response in patients treated with this regimen.
* Determine parameters that are associated with a high probability of response or non-response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive anti-thymocyte globulin IV over 8 hours on days 1-4. Patients also receive etanercept subcutaneously on days 8, 11, 15, and 18. Treatment with etanercept repeats every 28 days for at least 2 courses. Patients exhibiting hematologic improvement after course 2 may receive up to 2 additional courses of etanercept in the absence of disease progression or unacceptable toxicity. Patients with unresponsive disease or disease progression after course 2 are removed from the study and offered other treatment.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS)

  * Low- or intermediate-1-risk disease, as defined by International Prognostic Scoring System (IPSS) criteria, meeting 1 of the following criteria:

    * Single or multilineage cytopenia, as defined by all of the following:

      * Absolute neutrophil count < 1,500/mm^3
      * Hemoglobin < 10 g/dL
      * Platelet count < 100,000/mm^3
    * Transfusion requirement of ≥ 2 units of packed red blood cells within an 8-week period
* Not eligible for stem cell transplantation due to any of the following reasons:

  * No suitable bone marrow donor available
  * Not eligible for a transplantation protocol
  * Not willing to undergo transplantation
* No intermediate-2- or high-risk MDS
* No chronic myelomonocytic leukemia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No pneumonia within the past 2 weeks

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other severe disease that would preclude study compliance
* No other active severe infection (e.g., septicemia) within the past 2 weeks

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior and no concurrent hematopoietic growth factors for MDS
* More than 4 weeks since prior immunomodulatory therapy for MDS
* No prior anti-thymocyte globulin
* No prior hematopoietic stem cell transplantation
* No other concurrent immunomodulatory therapy for MDS

Chemotherapy

* Not specified

Endocrine therapy

* Prednisone < 5 mg/day allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since prior and no concurrent cytotoxic therapy for MDS
* More than 4 weeks since prior experimental therapy for MDS
* No other concurrent experimental therapy for MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Response rate
Correlate results of ex vivo/in vitro studies on phenotypic, cytogenetic, and functional disease characteristics with in vivo treatment responses
Identify parameters that are associated with a high probability of response

CONTACTS AND LOCATIONS:
Overall Officials: Bart L. Scott, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (4):
- United States (4):
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington